CLINICAL TRIAL: NCT02058108
Title: A Randomized, Double-blind, 104-weeks Treatment Study to Evaluate the Efficacy, Safety, Tolerability and Pharmacokinetics of Telbivudine Oral Solution and Tablets in Children and Adolescents With Compensated HBeAg-positive and Negative Chronic Hepatitis B Virus Infection
Brief Title: Study of Efficacy and Safety, Tolerability and Pharmacokinetics of Telbivudine in Children and Adolescents With Compensated Chronic Hepatitis B Virus Infection
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study terminated on the recommendation of an independent Data Monitoring Committee (DMC) subsequent to an interim efficacy analysis for futility.]
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CLDT600A2306; 2012-004942-14 (EudraCT Number)
Record Dates: First submitted 2014-02-05; First posted 2014-02-07 (Estimated); Results first posted 2019-09-10 (Actual); Last update posted 2019-09-10 (Actual); Status verified 2019-08

CONDITIONS: Chronic Hepatitis B
Keywords: Chronic hepatitis B, pediatrics, antiviral treatment, telbivudine
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — Telbivudine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Telbivudine (Experimental): Patients of any age and weight< 30kg: telbivudine oral solution (20 mg/mL): 20 mg/kg up to 600 mg q.d corresponding to weight (kg) x1mL, p.o. once daily Patients < 12 years old and weight≥ 30kg: telbivudine oral solution (20mg/mL), 600 mg/day corresponding to 30 mL p.o. once daily Patients ≥ 12 years old and weight ≥ 30kg: telbivudine film-coated tablet, 600 mg/day, corresponding to 1 tablet p.o. once daily
  Interventions: Drug: Telbivudine
- Placebo (Placebo Comparator): Patients of any age and weight < 30kg: placebo oral solution corresponding to weight (kg) x1mL, p.o. once daily Patients < 12 years old and weight ≥ 30kg: placebo oral solution corresponding to 30 mL p.o. once daily Patients ≥ 12 years old and weight ≥ 30kg: placebo tablet, corresponding to 1 tablet p.o. once daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Telbivudine — Patients of any age and weight< 30kg: telbivudine oral solution (20 mg/mL): 20 mg/kg up to 600 mg q.d corresponding to weight (kg) x1mL, p.o. once daily Patients < 12 years old and weight≥ 30kg: telbivudine oral solution (20mg/mL), 600 mg/day corresponding to 30 mL p.o. once daily Patients ≥ 12 years old and weight ≥ 30kg: telbivudine film-coated tablet, 600 mg/day, corresponding to 1 tablet p.o. once daily
  Arms: Telbivudine
Drug: Placebo — Patients of any age and weight < 30kg: placebo oral solution corresponding to weight (kg) x1mL, p.o. once daily Patients < 12 years old and weight ≥ 30kg: placebo oral solution corresponding to 30 mL p.o. once daily Patients ≥ 12 years old and weight ≥ 30kg: placebo tablet, corresponding to 1 tablet p.o. once daily
  Arms: Placebo

SUMMARY:
The purpose of the study was to assess the efficacy and safety of telbivudine at a dose of 20 mg/kg up to a maximum of 600 mg q.d. in compensated pediatric HBeAg-positive and negative CHB patients aged 2 to <18 years with the indication of antiviral CHB treatment. This study was part of the commitments of the pediatric development plan for telbivudine in Europe and US.

ELIGIBILITY:
Key Inclusion Criteria:

* Clinical history compatible with compensated chronic hepatitis B
* Documented compensated chronic hepatitis B defined by the following:

  1. Positive serum HBsAg at screening and at least one other documentation of HBsAg positive at least 6 months prior to screening
  2. For HBeAg positive patients at screening, significant biologic and/or histologic signs of disease activity following EASL guidelines recommendations for CHB pediatric patients (serum HBV DNA level ≥ 5 log10 copies/mL (or 20 000 IU/mL) (COBAS Taqman®) at screening ; serum ALT ≥ 1.5×ULN and < 10×ULN (pediatric ULN) for two times during the screening period or within 6 months prior to screening
  3. For HBeAg negative patients at screening, significant biologic and/or histologic signs of disease activity following EASL guidelines recommendations for CHB pediatric patients (serum HBV DNA level ≥ 4 log10 copies/mL (or 2 000 IU/mL) (COBAS Taqman®) at screening) ; serum ALT ≥ 1.0 ×ULN and < 10×ULN (pediatric ULN) for two times during the screening period or within 12 months prior to screening)

Key Exclusion Criteria:

* Patients with acute or chronic infection of HCV, HDV, HIV, or with acute infection of HAV, HEV, CMV, EBV, or HSV.
* Patient has received treatment of interferon or any other immunomodulatory agents within the last 12 months prior to screening or any nucleoside or nucleotide drugs or other anti-CHB treatment (approved or investigational) at any time before screening
* Patient has a medical condition that requires frequent use of systemic acyclovir or famciclovir, systemic corticosteroids, potentially hepatotoxic drugs or nephrotoxic drugs or chemotherapy
* Patient has one or more additional known primary or secondary causes of liver disease, other than CHB; has a decompensated liver disease ; is a Liver transplant recipient or organ or bone marrow transplant recipient.
* History of any other acute or chronic medical condition (that in the opinion of the investigator would make the patient unsuitable for inclusion into the study.
* Patient has a history of myopathy, myositis, persistent muscle weakness or persistent high serum CK levels (≥7×ULN), any muscular disease
* Patient receiving any drugs potentially associated with myopathy within 3 months prior to screening
* Any other clinical significant disease, condition or abnormality, unrelated to their HBV infection at screening, as assessed by the investigator

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 53 (Actual)
Dates: Start 2014-10-31 (Actual); Primary Completion 2019-01-09 (Actual); Study Completion 2019-01-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (26):
- Bulgaria (4):
  - Novartis Investigative Site, Sofia, Sofia-Grad
  - Novartis Investigative Site, Pleven
  - Novartis Investigative Site, Sofia
  - Novartis Investigative Site, Varna
- Greece (2):
  - Novartis Investigative Site, Goudi-Athens, GR
  - Novartis Investigative Site, Athens
- Israel (3):
  - Novartis Investigative Site, Jerusalem
  - Novartis Investigative Site, Nahariya
  - Novartis Investigative Site, Nazareth
- Romania (5):
  - Novartis Investigative Site, Cluj-Napoca, Cluj
  - Novartis Investigative Site, Craiova, Dolj
  - Novartis Investigative Site, Timișoara, Jud. Timis
  - Novartis Investigative Site, Bucharest
  - Novartis Investigative Site, Iași
- Novartis Investigative Site, Seoul, Korea, South Korea
- Turkey (Türkiye) (6):
  - Novartis Investigative Site, Ankara
  - Novartis Investigative Site, Antalya
  - Novartis Investigative Site, Diyarbakır
  - Novartis Investigative Site, Elâzığ
  - Novartis Investigative Site, Eskişehir
  - Novartis Investigative Site, Mersin
- Ukraine (5):
  - Novartis Investigative Site, Dnipropetrovsk
  - Novartis Investigative Site, Kiev
  - Novartis Investigative Site, Kyiv
  - Novartis Investigative Site, Odesa
  - Novartis Investigative Site, Vinnytsia

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted in 20 centers in 7 countries: Bulgaria (2), Greece (1), Israel (2), Republic of Korea (1), Romania (5), Turkey (4) and Ukraine (5 sites).
Pre-assignment Details: Patients were stratified by age group (2 to < 6 years, 6 to <12 years and 12 to <18 years) and HBV DNA level (low and high). At the baseline visit, eligible patients were randomized in a 24-week double blind period to telbivudine or placebo in a ratio 5:1. At Week 24 (visit 6), all patients were unblinded and HBV DNA level were assessed.
Groups:
- Placebo: Patients of any age and weight < 30kg: placebo oral solution corresponding to weight (kg) x1mL, p.o. once daily Patients < 12 years old and weight ≥ 30kg: placebo oral solution corresponding to 30 mL p.o. once daily Patients ≥ 12 years old and weight ≥ 30kg: placebo tablet, corresponding to 1 tablet p.o. once daily. Placebo randomized patients were offered optional telbivudine administration at week 24.
Period: Overall Study
Arm/Group | Telbivudine | Placebo
Started (All randomized patients were included in the Full Analysis (FAS) and Safety Set) | 43 | 10
Switched to Telbivudine After Week 24 (Placebo randomized patients who switched to LdT after week 24) | 0 | 5
Completed | 2 | 0
Not Completed | 41 | 10
Not completed — Abnormal Laboratory Values | 0 | 1
Not completed — Unsatisfactory therapeutic effect | 37 | 4
Not completed — No longer requires study drug | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Administrative problems | 3 | 3
Not completed — Protocol Violation | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Telbivudine | Placebo | Total
Number analyzed (Participants) | 43 | 10 | 53
Age, Continuous [Mean (Standard Deviation); unit: Years] | 10.2 (4.88) | 9.1 (4.89) | 10.0 (4.86)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 4 | 18
  Male | 29 | 6 | 35
Race/Ethnicity, Customized [Number; unit: Participants]
  Caucasian | 40 | 10 | 50
  Black | 1 | 0 | 1
  Asian | 2 | 0 | 2
HBV DNA [Mean (Standard Deviation); unit: log10 copies/mL] | 9.1 (1.14) | 8.2 (2.26) | 8.9 (1.43)
Participants with alanine aminotransferase (ALT) - Multiples of upper limits of normal (ULN) [Count of Participants; unit: Participants] — Serum ALT normalization is an important clinically relevant efficacy endpoint. Elevated serum ALT levels are thought to reflect underlying hepatitis disease activity (i.e. active liver inflammation). Correspondingly, ALT normalization is an accepted therapeutic goal in hepatitis studies as it is thought to reflect a substantial reduction in hepatic disease activity. Measurement at baseline.
  Participants
    < 1 × ULN | 4 | 3 | 7
    1 × - < 2 × ULN | 22 | 4 | 26
    2 × - < 5 × ULN | 16 | 2 | 18
    5 × or more ULN | 1 | 1 | 2
Participants with aspartate aminotransferase (AST) - Multiples of upper limits of normal (ULN) [Count of Participants; unit: Participants]
  < 1 × ULN | 26 | 5 | 31
  1 × - < 2 × ULN | 14 | 4 | 18
  2 × - < 5 × ULN | 2 | 0 | 2
  5 × or more ULN | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Achieving Serum HBV DNA Level of <300 Copies/mL (51 IU/mL) at Week 24
Description: The primary objective of this study was to demonstrate the antiviral efficacy of telbivudine compared to placebo in pediatric patients (2- < 18 years) by determining the percentage of patients achieving serum HBV DNA level of <300 copies/mL (51 IU/mL) at Week 24.
Time Frame: Week 24
Population: The Full Analysis Set (FAS), which consisted of all randomized patients to whom study treatment had been assigned, was considered.
Measure: Count of Participants; unit: Participants
Arm/Group | Telbivudine | Placebo
Number analyzed (Participants) | 41 | 8
Participants | 5 | 1
Statistical Analysis 1: Comparison: Telbivudine vs Placebo; HBV DNA level of <300 copies/mL (51 IU/mL) at Week 24; Test type: Other — Missing assessment imputed using the closest available assessment; p = 1.0000, Fisher Exact; Mean Difference (Net) = -0.30, 95% CI 2-sided [-37.03 to 36.75]; Exact confidence interval for the difference in percentage

2. Secondary Outcome: Number of Patients Achieving HBV DNA< 300 Copies/mL (51 IU/mL) at Week 52 and Week 104
Description: The antiviral efficacy at Weeks 52 and 104 was to be evaluated by: a) the proportion of patients achieving HBV DNA <300 copies/mL (51 IU/mL) at Week 52 and Week 104; b) the proportion of patients achieving HBV DNA < Lower Limit of Quantification (LLOQ), <1000 copies/ml (or 200 IU/mL), <10,000 copies/ml (or 2 000 IU/mL) and ≥10,000 copies/mL (or 2 000 IU/mL) at Week 24, 52 and 104; c) the proportion of patients achieving Serum HBV DNA reduction from baseline; d) the time to achieve HBV DNA <300 copies/mL (51 IU/mL); e) the proportion of patients with Primary non-response.
  Due to early termination of the study and limited number of enrolled patients on track to complete 52 weeks of participation (8 patients overall), only descriptive analysis performed at Week 52 and Week 104.
Time Frame: Week 52, Week 104
Population: The Full Analysis Set (FAS), which consisted of all randomized patients to whom study treatment had been assigned, was considered. Only patients with efficacy data within censoring date included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Telbivudine | Placebo
Number analyzed (Participants) | 3 | 3
Participants
  Week 52 | 3 | 0
  Week 104: number analyzed (Participants) | 2 | 0
  Week 104 | 2 |

3. Secondary Outcome: Number of Patients Whose Baseline ALTs Were Abnormal and Subsequently Normalized at Week 24, 52 and 104
Description: The biochemical response at Weeks 24, 52 and 104 was to be evaluated by the proportion of patients whose baseline ALTs were abnormal (defined as ALT >1 x Upper Limit of Normal [ULN]) and subsequently normalized.
  Due to early termination of the study and limited number of enrolled patients on track to complete 52 weeks of participation (8 patients overall), only descriptive analysis performed at Week 52 and Week 104.
Time Frame: Week 24, Week 52, Week 104
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Telbivudine | Placebo
Number analyzed (Participants) | 37 | 5
Participants
  Week 24 | 12 | 0
  Week 52: number analyzed (Participants) | 3 | 3
  Week 52 | 1 | 1
  Week 104: number analyzed (Participants) | 2 | 0
  Week 104 | 2 |
Statistical Analysis 1: Comparison: Telbivudine vs Placebo; ALT levels at Week 24; Test type: Other; p = 0.2984, Fisher Exact; Mean Difference (Net) = 32.43, 95% CI 2-sided [-14.62 to 74.60] — Exact confidence interval for the difference in percentage. P-value from Fishers exact test comparing proportions in Initial LdT and Initial Placebo groups

4. Secondary Outcome: Number of Patients With HBeAg Loss, HBeAg Seroconversion at Week 24, 52 and 104
Description: The serological response at Weeks 24, 52 and 104 was to be evaluated by: a) the proportion of HBeAg positive patients at baseline who subsequently have HBeAg loss and HBeAg seroconversion (defined as loss of HBeAg with detectable HBeAb); b) the proportion of HBsAg positive patients at baseline who subsequently have HBsAg loss and HBsAg seroconversion (defined as loss of HBsAg with detectable HBsAb).
  Due to early termination of the study and limited number of enrolled patients on track to complete 52 weeks of participation (8 patients overall), only descriptive analysis performed at Week 52 and Week 104.
Time Frame: Week 24, Week 52, Week 104
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Telbivudine | Placebo
Number analyzed (Participants) | 37 | 4
Participants
  HBeAg loss at Week 24 | 1 | 0
  HBeAg seroconversion at Week 24 | 1 | 0
  HBeAg loss at Week 52: number analyzed (Participants) | 3 | 3
  HBeAg loss at Week 52 | 1 | 0
  HBeAg seroconversion at Week 52: number analyzed (Participants) | 3 | 3
  HBeAg seroconversion at Week 52 | 1 | 0
  HBeAg loss at Week 104: number analyzed (Participants) | 2 | 0
  HBeAg loss at Week 104 | 1 |
  HBeAg seroconversion at Week 104: number analyzed (Participants) | 2 | 0
  HBeAg seroconversion at Week 104 | 1 |
Statistical Analysis 1: Comparison: Telbivudine vs Placebo; HBeAg loss at Week 24; Test type: Other; p = 1.0000, Fisher Exact; Mean Difference (Net) = 2.70, 95% CI 2-sided [-53.70 to 60.20] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 2: Comparison: Telbivudine vs Placebo; HBeAg seroconversion at Week 24; Test type: Other; p = 1.0000, Fisher Exact; Mean Difference (Net) = 2.70, 95% CI 2-sided [-53.70 to 60.20] — [estimate comment as in outcome 3, analysis 1]

5. Secondary Outcome: Number of Patients With HBsAg Loss, HBsAg Seroconversion at Week 24, 52 and 104
Description: as for outcome 4
Time Frame: Week 24, Week 52, Week 104
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Telbivudine | Placebo
Number analyzed (Participants) | 41 | 7
Participants
  HBsAg loss at Week 24 | 1 | 0
  HBsAg seroconversion at Week 24 | 0 | 0
  HBsAg loss at Week 52: number analyzed (Participants) | 3 | 3
  HBsAg loss at Week 52 | 0 | 0
  HBsAg seroconversion at Week 52: number analyzed (Participants) | 3 | 3
  HBsAg seroconversion at Week 52 | 0 | 0
  HBsAg loss at Week 104: number analyzed (Participants) | 2 | 0
  HBsAg loss at Week 104 | 0 |
  HBsAg seroconversion at Week 104: number analyzed (Participants) | 2 | 0
  HBsAg seroconversion at Week 104 | 0 |
Statistical Analysis 1: Comparison: Telbivudine vs Placebo; HBsAg loss at Week 24; Test type: Other; p = 1.0000, Fisher Exact; Mean Difference (Net) = 2.44, 95% CI 2-sided [-37.54 to 42.17] — [estimate comment as in outcome 3, analysis 1]

6. Secondary Outcome: Number of Patients Achieving a Composite Endpoints (HBV DNA < 300 Copies/mL (51 IU/mL), ALT Normalization and HBeAg Seroconversion) at Week 52 and 104
Description: The proportion of patients achieving composite endpoints at Week 52 and 104 was to be evaluated by the proportion of patients achieving: a) HBV DNA <300 copies/mL (51 IU/mL); b) ALT normalization and HBeAg seroconversion for HBeAg positive patients only; c) HBV DNA <300 copies/mL (51 IU/mL) and ALT normalization for HBeAg negative patients.
  Due to early termination of the study and limited number of enrolled patients on track to complete 52 weeks of participation (8 patients overall), only descriptive analysis performed at Week 52 and Week 104.
Time Frame: Week 52, Week 104
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Telbivudine | Placebo
Number analyzed (Participants) | 3 | 3
Participants
  Week 52 | 1 | 0
  Week 104: number analyzed (Participants) | 2 | 0
  Week 104 | 1 |

7. Secondary Outcome: Number of Patients Achieving Cumulative Rate of Virological Breakthrough (VB) at Week 52 and 104
Description: The assessment of virological breakthrough (VB) was to be evaluated by: a) the cumulative rate of patients with confirmed VB at Week 52 and Week 104; b) the time to VB.
  Due to early termination of the study and limited number of enrolled patients on track to complete 52 weeks of participation (8 patients overall), only descriptive analysis performed at Week 52 and Week 104.
Time Frame: Week 52, Week 104
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Telbivudine | Placebo
Number analyzed (Participants) | 41 | 8
Participants
  Week 52 | 1 | 0
  Week 104 | 1 | 0

8. Secondary Outcome: Number of Participants With Treatment Emergent Genotypic Resistance Associated With VB, or in Patients With HBV DNA≥300 Copies/mL (51 IU/mL) at Week 24 and Discontinued From the Study
Description: Assessment of the presence of treatment emergent genotypic resistance (confirmed by genotypic sequencing) associated with virological breakthrough over the study period, or in patients with HBV DNA≥300 copies/mL (51 IU/mL) at Week 24 and discontinued from the study treatment (or at discontinuation if prior to Week 24 for subjects with at least 16 weeks of LDT treatment)
Time Frame: Week 24
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Telbivudine | Placebo
Number analyzed (Participants) | 41 | 8
Participants
  Cumulative virological breakthrough | 0 | 0
  Cumulative treatment emergent genotypic resistance: number analyzed (Participants) | 40 | 7
  Cumulative treatment emergent genotypic resistance | 1 | 0
Statistical Analysis 1: Comparison: Telbivudine vs Placebo; Treatment emergent genotypic resistance at Week 24; Test type: Other; p = 1.0000, Fisher Exact; Mean Difference (Net) = 2.50, 95% CI 2-sided [-37.05 to 41.83] — [estimate comment as in outcome 3, analysis 1]

9. Secondary Outcome: Number of Participants With On-Treatments Adverse Events, Serious Adverse Events, and Death
Description: Evaluation of the safety and tolerability of Telbivudine defined by AEs, SAEs, adverse events of special interest (AESI) (including muscle related events) and death; laboratory evaluations specifically on-treatment and post-treatment ALT flares, incidence and clinical significance of CK elevations; growth and development (linear growth and sexual maturation); development of liver decompensation and/or HCC.
  Only descriptive analysis performed.
Time Frame: From first dose of study treatment to 30 days after last dose of study treatment, up to 112 weeks
Population: The Safety Set, which consisted of all patients who received at least one dose of study drug during the treatment period, was considered.
Measure: Count of Participants; unit: Participants
Arm/Group | Telbivudine | Placebo
Number analyzed (Participants) | 43 | 10
Participants
  On-treatment Adverse Event (AEs) | 20 | 4
  On-treatment Serious Adverse Event (SAEs) | 0 | 0
  On-treatment Deaths | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events and serious adverse events were collected for the maximum actual duration of treatment exposure and follow up for a participant per the protocol for approximately 112 weeks.
Description: Adverse events occurring in patients in the Initial Placebo group were assigned to either Placebo or Telbivudine (LdT) treatment based on their onset date:
  * Placebo: AEs with onset before the first date of LdT treatment after switching; for patients who did not switch to LdT, all AEs were assigned to Placebo
  * LdT: AEs with onset date on or after the first date of LdT treatment after switching.
Groups:
- Initial LdT (Telbivudine): Patients of any age and weight< 30kg: telbivudine oral solution (20 mg/mL): 20 mg/kg up to 600 mg q.d corresponding to weight (kg) x1mL, p.o. once daily Patients < 12 years old and weight≥ 30kg: telbivudine oral solution (20mg/mL), 600 mg/day corresponding to 30 mL p.o. once daily Patients ≥ 12 years old and weight ≥ 30kg: telbivudine film-coated tablet, 600 mg/day, corresponding to 1 tablet p.o. once daily
- Initial Placebo on Placebo Treatment: Initial Placebo patients who did not switched to LdT treatment
- Initial Placebo on LdT Treatment After Switching: Initial Placebo patients who switched to LdT treatment
- All Ldt: Initial LdT and Initial Placebo on LdT treatment after switching combined
Arm/Group | Initial LdT (Telbivudine) | Initial Placebo on Placebo Treatment | Initial Placebo on LdT Treatment After Switching | All Ldt
All-Cause Mortality (participants affected / at risk) | 0/43 | 0/10 | 0/5 | 0/48
Serious Adverse Events (participants affected / at risk) | 0/43 | 0/10 | 0/5 | 0/48
Other Adverse Events (participants affected / at risk) | 20/43 | 4/10 | 1/5 | 21/48
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Initial LdT (Telbivudine) (N=43) | Initial Placebo on Placebo Treatment (N=10) | Initial Placebo on LdT Treatment After Switching (N=5) | All Ldt (N=48)
Ear pain (Ear and labyrinth disorders) | 0 | 1 | 0 | 0
Conjunctival hyperaemia (Eye disorders) | 1 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 5 | 0 | 0 | 5
Diarrhoea (Gastrointestinal disorders) | 2 | 0 | 0 | 2
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Exanthema subitum (Infections and infestations) | 1 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 2 | 0 | 0 | 2
Laryngitis (Infections and infestations) | 1 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 0 | 1 | 1
Otitis media (Infections and infestations) | 1 | 0 | 0 | 1
Pharyngitis (Infections and infestations) | 1 | 0 | 0 | 1
Tonsillitis (Infections and infestations) | 1 | 1 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 1 | 0 | 1
Varicella (Infections and infestations) | 1 | 0 | 0 | 1
Viral infection (Infections and infestations) | 1 | 0 | 0 | 1
Viral upper respiratory tract infection (Infections and infestations) | 3 | 0 | 0 | 3
Blood creatine phosphokinase increased (Investigations) | 2 | 0 | 0 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 1
Headache (Nervous system disorders) | 6 | 1 | 0 | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 2
Antibiotic prophylaxis (Surgical and medical procedures) | 0 | 1 | 0 | 0

LIMITATIONS AND CAVEATS:
Due to early termination of the study and limited number of enrolled patients on track to complete 52 weeks of participation (8 patients overall), no formal analysis of Weeks 52 and 104 long-term efficacy endpoints (only descriptive analysis).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2016-11-22): https://cdn.clinicaltrials.gov/large-docs/08/NCT02058108/Prot_000.pdf
  • Statistical Analysis Plan (2017-09-25): https://cdn.clinicaltrials.gov/large-docs/08/NCT02058108/SAP_001.pdf